CLINICAL TRIAL: NCT00291304
Title: Magnetic Resonance Imaging (MRI) Correlation to Standard of Care Imaging and Pathology Correlation in Breast Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BR-1-0082
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
Keywords: Magnetic Resonance Imaging; Pathology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MRI — pre-surgery

SUMMARY:
Magnetic Resonance Imaging (MRI) is a well known imaging tool for the investigation and diagnosis of breast cancer, used in addition to breast mammograms and ultrasound. Recent publications suggest that MRI may be the best test to use in women who have very dense breasts, have a family history of breast cancer and have had breast cancer and were treated with breast saving measures. MRI has been shown to be a better tool to show multiple breast cancer spots than mammography or ultrasound. The radiologists and the radiology students will have the opportunity to review the MRI scans along with the breast ultrasound and mammography films and the pathology reports from the breast cancer surgery completed at the CCI. This may enable them to learn how the various subtypes of breast cancer look on MRI. The goal is: 1) to gain good breast MRI expertise, giving the Radiology residents a complete diagnostic program. 2) to develop good MRI breast experience, enabling the Cross Cancer Institute to be the centre of excellence for Breast MRI for northern Alberta.

DETAILED DESCRIPTION:
Background Information

In addition to the gold standard imaging of mammography and breast ultrasound, magnetic resonance imaging (MRI) has become a well established investigational modality for the diagnosis and staging of breast cancer. MRI demonstrates increased sensitivity and specificity relative to both mammography and breast ultrasound in the screening of women with an increased risk of breast cancer development (i.e. familial history of disease and / or genetic predisposition) and those who have very dense breast tissue. MRI has also proved to be very sensitive in the detection of multi-focal, multi-centric breast lesions, permitting the accurate staging of disease. However, despite this demonstrated efficacy, the standardization of MRI studies from one Institution to another is often difficult as each Institution will have a standard breast protocol with sequences set in accordance to the manufacturer of the machine and the manner in which the breast examinations have been designed.

At the Cross Cancer Institute (CCI) a breast MRI protocol based on the technical procedures recommended in the literature and personal scanning experience has been developed. However, due to the limited number of patients undergoing breast MRI examinations, our current experience is limited relative to the level of expertise demonstrated in the interpretation of breast ultrasound and mammographic scans. Fortunately, we now have the opportunity to obtain MRI - pathology correlation as Dr. Kelly Dabbs is performing on site breast cancer surgery at the CCI. We propose to obtain an MRI examination of all consented patients prior to their surgical procedure. The MRI results of each patient will then be compared to previous breast imaging (mammography and breast ultrasound) and histopathological specimens to determine the correlative accuracy of MRI with these techniques. To assess whether the size, grade, and presence of lymphovascular invasion or associated ductal carcinoma in situ influence the accuracy of MR imaging, all breast carcinoma subtypes will be included in this study.

As a teaching hospital, the CCI provides mammographic and breast ultrasound training to the Residents and the Diagnostic Radiology Program at the University of Alberta. Although breast MRI should be part of this training program, we currently do not have the necessary volume of breast MRI scans to provide Residents with adequate experience in this modality. The establishment of a breast MRI protocol, one which refers eligible CCI breast cancer patients for a pre-surgery MRI examination, will promote the development of expertise in this area, provide Residents with a comprehensive Breast program and keep the CCI at the leading edge of breast cancer care.

Objectives

Primary Objective: to assess how the MRI of the breast correlates to a standard of care which includes biopsy, surgery, breast ultrasound and mammography.

Secondary Objective: to assess how the MRI correlates to the breast cancer pathology collected at the CCI.

Study Design

A research study is proposed with the above information in mind, whereby Dr. Kelly Dabbs refers consented surgical patients with known breast carcinoma for a pre-surgical breast MRI. The MRI results will then be reviewed along with the mammograms and breast ultrasounds and then correlated to pathology findings. The intent will be to correlate all of the various sub-types of breast carcinoma with MRI, as well as to assess whether or not MRI demonstrates changes dependent upon the extent lymphovascular invasion, the presence of associated ductal carcinoma in situ and the size, cellular composition and grade of the cancer.

Dr. Dabbs will explain the study rational and give the patient a copy of Informed Consent and, for those patients who are willing to undergo the procedure, schedule a MRI at the CCI. It is our aim to accrue 50 patients per year for two years, for a total of 100 patients.

Inclusion / Exclusion Criteria

Inclusion criteria:

* Females ? 18 years of age
* Females referred to Dr. Kelly Dabbs for breast cancer surgery who have pathology positive for breast carcinoma, any sub-type.

Exclusion criteria:

* Pacemakers
* Aneurysm clips
* Cochlear implants
* Epicardial pacemaker wires
* Neural stimulators
* Significant claustrophobia
* Significant obesity that would not enable the patient to fit in the scanner
* Pregnancy or breastfeeding

Recruitment

Surgical patients referred by Dr. Kelly Dabbs will undergo a pre-surgical MRI examination providing they meet the study eligibility criteria.

Statistical analysis

N/AP

Stopping Rules

The study will end once the first 100 subjects enrolled have undergone their MRI breast scan.

Data Safety Monitoring Committee

N/AP

ELIGIBILITY:
Inclusion Criteria:

* females 18 years or older
* females referred to Dr. Kelly Dabbs for breast cancer surgery with pathology positive for breast carcinoma, any subtype

Exclusion Criteria:

* pacemakers
* aneurysm clips
* cochlear implants
* epicardial pacemaker wires
* neural stimulators, etc.
* significant claustrophobia
* significant obesity that would not enable the patient to fit in the scanner
* pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
-assess how MRI of the breast correlates to standard of care which includes ultrasound, mammography, biopsy and surgery | 2 years

SECONDARY OUTCOMES:
-assess how the MRO correlates to the breast cancer pathology collected at the CCI | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Campbell, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada